CLINICAL TRIAL: NCT04414358
Title: Incidence of Residual Significant Tricuspid Regurgitation in Patients Undergoing Left-sided Cardiac Surgery
Brief Title: Incidence of Residual Tricuspid Regurgitation in Patients Undergoing Left-heart Surgery
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-3
Record Dates: First submitted 2020-05-31; First posted 2020-06-04 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Residual Tricuspid Regurgitation; Left-sided Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Functional tricuspid valve regurgitation is commonly co-existed with left-sided cardiac lesion, especially mitral valve stenosis. Both lesion were recommended to surgically fixed at the same setting. Residual tricuspid regurgitation may effects patients' outcome. The investigators would like to determine the incidence of significant residual tricuspid regurgitation after left-sided cardiac surgery and related clinical outcome.

DETAILED DESCRIPTION:
Functional tricuspid regurgitation (TR) was defined as TR occurring secondary to left heart, especially mitral valve stenosis or pulmonary disease. Previous study reported that about 30% - 50% of patients with significant mitral stenosis developed moderate to severe TR. In the past, corrective TR repair was not always indicated because the concept about TR severity will improve after mitral valve lesion was treated.

Later on, several studies demonstrated that the patients with untreated significant (< moderate) TR had worse clinical outcome including mortality. While simultaneous functional TR repair with left-sided valve surgery did not cause adverse events, but improve clinical outcome and quality of life. The current European Society of Cardiology (ESC)/European Association for Cardio-Thoracic Surgery (EACTS) and American Heart Association(AHA)/American College of Cardiology (ACC) guidelines recommend concomitant tricuspid valve (TV) surgery in patients with severe TR undergoing left-sided valve surgery (class I recommendation). In patients with mild to moderate TR, there is a class IIa indication for concomitant TV surgery in the setting of tricuspid annular dilatation.

However, after TV repair, commonly with annuloplasty ring or De Vega annuloplasty, residual TR may still persist and the residual moderate or severe TR have negative impact to right ventricle (RV). It can cause RV dilatation and RV failure(7, 12). Calafiore et al reported 12.4% of significant TR after surgery and the associated factors for the repair failure. If this group of patients developed symptom of RV failure or progressive RV dilatation or dysfunction is detected, they possessed very high-risk for re-operation.

Preoperative transthoracic echocardiography (TTE) is an important tool to classified severity of TR, measured TV annulus, indicate the surgical correction requirement and demonstrate the result of the TR repair. Due to limitation of TTE operator and machine, time-interval between the latest preoperative TTE result and surgery are varied, so the TR severity may already changed. The postoperative TTE result sometimes comes out late after surgery. Therefore, transesophageal echocardiography (TEE), operated by trained cardiac anesthesiologist, may play role to confirm the severity and provide the instant result of the TV repair to help guide the cardiac surgeon to make a decision whether to re-operate in the same setting to improve the surgical outcome.

Therefore, the investigators would like to determine the incidence of residual significant TR by intraoperative TEE in the patients underwent left-side cardiac surgery and the related clinical outcome, including rate of re-admission from cardiac cause and 1- year mortality.

ELIGIBILITY:
Inclusion Criteria:

* Mitral valve or aortic valve diseases requiring surgical intervention
* No pathologic changes in TV leaflets
* No previous tricuspid valve surgery

Exclusion Criteria:

* Patients with incomplete data
* Patient with history of previous cardiac surgery
* Patient with congenital anomalies of mitral or tricuspid valve
* Patient with both tricuspid stenosis and regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients scheduled for surgery according to the criteria in Siriraj hospital, Mahidol university will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with residual significant tricuspid regurgitation after left-sided cardiac surgery | during surgery
  * Residual significant tricuspid regurgitation: more than moderate tricuspid regurgitation after corrective surgery
  * Left-sided cardiac surgery: mitral or aortic valve surgery

SECONDARY OUTCOMES:
Number of patients with different severity of tricuspid regurgitation | during surgery
  Compare between preoperative trans- thoracic echocardiography and intraoperative transesophageal echocardiography result (before cardiopulmonary bypass initiation)
Length of stay | 7 days after surgery
  Length of hospital and ICU stay
Number of patients require re-operation | 1 year after surgery
  Re-operation for tricuspid regurgitation correction
Number of patients require re-admission | 1 year after surgery
  Re-admission due to cardiac cause: right-sided cardiac failure, pulmonary oedema

CONTACTS AND LOCATIONS:
Overall Officials: Aphichat Suphathamwit, M.D>, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anyanwu AC, Adams DH. Functional tricuspid regurgitation in mitral valve disease: epidemiology and prognostic implications. Semin Thorac Cardiovasc Surg. 2010 Spring;22(1):69-75. doi: 10.1053/j.semtcvs.2010.05.006. PMID 20813320
- [Background] Hamandi M, George TJ, Smith RL, Mack MJ. Current outcomes of tricuspid valve surgery. Prog Cardiovasc Dis. 2019 Nov-Dec;62(6):463-466. doi: 10.1016/j.pcad.2019.11.014. Epub 2019 Dec 2. PMID 31805294
- [Background] Calafiore AM, Foschi M, Kheirallah H, Alsaied MM, Alfonso JJ, Tancredi F, Gaudino M, Di Mauro M. Early failure of tricuspid annuloplasty. Should we repair the tricuspid valve at an earlier stage? The role of right ventricle and tricuspid apparatus. J Card Surg. 2019 Jun;34(6):404-411. doi: 10.1111/jocs.14042. Epub 2019 Apr 8. PMID 30958905